CLINICAL TRIAL: NCT00315107
Title: Estrogen Treatment in Acromegalic Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HND01
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2006-05

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Ethinyl Estradiol-Norgestrel Combination

INTERVENTIONS:
Drug: Alesse

SUMMARY:
Oral estrogens may be an effective adjuvant treatment for control of acromegaly in patients with resistance to somatostatin analogs.

DETAILED DESCRIPTION:
This will be a canadian multicenter study with a randomized, double-blind, placebo-controlled design, to assess the efficacy and safety of adjuvant alesse in female acromegalic patients with suboptimal response to sandostatin LAR treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older treated with somatostatin analogs
* Active acromegaly

Exclusion Criteria:

* Cardiovascular or cerebrovascular disease
* Thrombophlebitis or thromboembolism
* Breast cancer
* Non-controlled arterial hypertension
* Smoking
* Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-05; Study Completion 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Omar Serri, MD, Principal Investigator — CHUM- Endocrinology
Locations (1):
- CHUM - Notre-Dame Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Kestler E, Ambrosio G, Hemming K, Hughes JP, Matute J, Moreno M, Madriz S, Walker D. An integrated approach to improve maternal and perinatal outcomes in rural Guatemala: A stepped-wedge cluster randomized trial. Int J Gynaecol Obstet. 2020 Oct;151(1):109-116. doi: 10.1002/ijgo.13262. Epub 2020 Jul 27. PMID 32524605